CLINICAL TRIAL: NCT00641108
Title: Effect of Psychotherapy on Brain Serotonin Activity
Brief Title: Effects of Cognitive Behavioral Therapy on Brain Serotonin Activity in People With Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R34MH077580 (NIH); R34MH077580 (NIH); DATR A5-ETMA
Record Dates: First submitted 2008-03-19; First posted 2008-03-21 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Depression
Keywords: SPECT Brain Imaging; Cognitive Therapy; Serotonin Transporter Binding; Predictive Biomarker
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADAM SPECT (Experimental): Participants with depression will undergo ADAM SPECT scans and cognitive behavioral therapy.
  Interventions: Drug: ADAM SPECT plus Cognitive Therapy
- Control (Active Comparator): Healthy subjects without depression will undergo ADAM SPECT scans.
  Interventions: Drug: ADAM SPECT plus No Therapy

INTERVENTIONS:
Drug: ADAM SPECT plus Cognitive Therapy
  Arms: ADAM SPECT
Drug: ADAM SPECT plus No Therapy
  Arms: Control

SUMMARY:
This study will examine changes in brain serotonin activity in people with depression before and after they receive cognitive behavioral therapy.

DETAILED DESCRIPTION:
Depression is a serious illness that affects almost 19 million adults in the United States each year. Common symptoms of depression include persistent feelings of anxiety, guilt, or hopelessness; irregular sleep and appetite patterns; lethargy; disinterest in previously enjoyed activities; excessive irritability and restlessness; suicidal thoughts; and inability to concentrate. A person's depression can be attributed to a variety of causes, including biological and genetic factors, environmental influences, or developmental experiences. Among biological factors, a recently researched possible cause is the altered activity of specialized areas on brain nerve cells called serotonin receptors, which have been found to be at reduced levels in people with depression. The hormone serotonin is known to naturally influence mood, making depression treatments that aim to increase levels of serotonin important. Treatment for depression with cognitive behavioral therapy (CBT), which teaches ways to modify thoughts and behaviors that contribute to depression, may help in raising brain serotonin levels and in improving depressive symptoms. This study will examine changes in brain serotonin activity using single photon emission computed tomography (SPECT) imaging in people with depression before and after they receive CBT. The study will also use SPECT imaging to compare brain serotonin activity of non-depressed healthy participants with that of depressed participants.

Participation in this study will last between 12 and 14 weeks. All participants will first undergo an initial evaluation that will include questions about medical history, a physical exam, a blood draw, a urine test, and an electrocardiogram (ECG). Participants will then undergo an ADAM (a selective radioligand for SPECT imaging) SPECT scan. During the ADAM SPECT scan visit, participants will undergo an injection of the ADAM, an ECG, blood pressure monitoring, and a 60-minute SPECT scan. If necessary, participants may also be asked to have a magnetic resonance imaging (MRI) brain scan after completing the SPECT scan.

Depressed participants will then attend at least once weekly CBT sessions for 12 weeks. During the 45-minute sessions, participants will meet with a therapist to learn ways to adjust thoughts and behaviors that may be adding to their depression. After completing the 12 weeks of CBT, all participants will be re-evaluated by a study doctor and, if still in good health, will undergo a repeat ADAM SPECT scan.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depressive disorder (MDD)
* Drug naive from prior psychotropic medication for more than 6 months before study entry
* Hamilton-Depression (HAM-D) 17 score greater than or equal to 16
* Woman of childbearing age with a negative pregnancy test within 48 hours of scanning

Exclusion Criteria:

* DSM-IV Axis I diagnosis other than MDD
* Use of psychotropic medication within 6 months of study entry
* History of bipolar disorder
* Current alcohol or drug abuse/dependence within 6 months of study entry
* History of sensitivity or intolerance to s-citalopram
* Medical contraindication to the use of s-citalopram
* Unstable medical condition (e.g., angina pectoris, untreated hypertension)
* Pregnant or nursing
* Woman of childbearing potential not using a medically acceptable form of birth control
* Actively suicidal or requiring hospitalization
* Requiring additional psychotropic drug therapy
* History of transient ischemic attacks
* History of cerebral infarction (including lacunar infarct with symptoms more than 24 hours in duration)
* History of Binswanger's disease or a history of hypertensive encephalopathy
* History of intracranial hemorrhage
* History of head trauma with loss of consciousness
* History of encephalitis
* History of extended exposure to known neurotoxin (e.g., cyanide, carbon monoxide)
* Uncontrolled metabolic disorder (e.g., thyroid disease, diabetes mellitus)
* History of cognitive impairment other than major depressive episode
* History of normal pressure hydrocephalus
* History of cancer metastatic to the central nervous system
* History of Parkinson's or other basal ganglia disease
* History of Guillain-Barré syndrome (chronic or relapsing polyneuropathy)
* Inability to undergo an MRI scan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. DeRubeis, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit - University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Groups:
- ADAM SPECT: Participants with depression will undergo ADAM SPECT scans and cognitive behavioral therapy.
  ADAM SPECT plus Cognitive Therapy
- Control: Healthy subjects without depression will undergo ADAM SPECT scans.
  ADAM SPECT plus No Therapy
Period: Overall Study
Arm/Group | ADAM SPECT | Control
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Groups:
- Total: Total of all reporting groups
Arm/Group | ADAM SPECT | Control | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized [unit: participants]
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Serotonin Transporter Availability
Time Frame: Measured at Weeks 0 and 12
Population: as for baseline characteristics
Arm/Group | ADAM SPECT | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Arm/Group | ADAM SPECT | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data is unavailable due to the following extenuating circumstances: principal investigator has serious health complications preventing him from inputting data, and study team has left university and is unreachable to input data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes